CLINICAL TRIAL: NCT05195307
Title: Effectiveness of Music Therapy on Anxiety and Stress Levels of Primiparous Pregnants in the Third Trimester: A Randomised Controlled Trial
Brief Title: The Effect of Music Therapy Applied to Pregnant Women on Anxiety and Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Ebru Ertas, Research Assistant, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Ayşe Koçak Sezgin
Record Dates: First submitted 2021-12-15; First posted 2022-01-18 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Music Therapy
Keywords: midwifery; pregnancy; music; anxiety; stress
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: A randomized study with an application and a control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Group (Experimental): Application Group Pregnant women in the application group were regularly listened to music for 20 minutes a day for 10 days. In addition, the pregnant women in the application group were trained by the researcher on preparing for normal delivery.
  Interventions: Other: Music Group
- Control Group (No Intervention): In the study, pregnant women in the control group were trained by the researcher on preparing for normal delivery.

INTERVENTIONS:
Other: Music Group — Pregnant women included in the practice group were given 20 minutes of music every day for ten days. Anxiety and stress levels of pregnant women were measured before and after the intervention.
  Arms: Music Group

SUMMARY:
Anxiety and stress increase in primiparous pregnant women and especially in the third trimester of pregnancy. This study was conducted to investigate the effect of music therapy applied to pregnant women who will give birth for the first time and are in the last trimester of their pregnancy on anxiety and stress. The study is a randomized controlled trial. Pregnant women in the application group were regularly listened to music for 20 minutes a day for 10 days. In the study, pregnant women in the application and control group were trained by the researcher on preparing for normal delivery. The pregnant women who participated in the study completed the Personal Information Form, the State and Trait Anxiety Inventory and the Pregnancy Stress Rating Scale at the beginning. 10, the last day of study. on the day, the scales are repeated.

DETAILED DESCRIPTION:
Aims and objectives: This study aimed to evaluate the effect of music therapy on the anxiety and stress levels of primiparous pregnants in the third trimester.

Background: Anxiety and stress during pregnancy, when not well-managed, can lead to negative birth outcomes.

Design: This study is a randomized controlled trial. Methods: This study was conducted in Turkey with 120 pregnant, 60 of whom were in the music group and 60 in the control group. Research data were collected with Personal Information Form, State-Trait Anxiety Inventory and Pregnancy Stress Rating Scale-36. Pregnants were made to listen to music for 20 minutes every day for ten days. The anxiety and stress levels of pregnant were measured before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 18 and over,
* Primiparous pregnants,
* In the third trimester (28 and above gestational week),
* Speaking and writing in Turkish,
* Having no vision-hearing problems,
* Having and using internet-supported online Web 2.0 tools,
* Volunteering to participate in the study were included in the study within the scope of inclusion criteria.

Exclusion Criteria:

* Pregnant women who did not meet the inclusion criteria and pregnant women who did not listen to music regularly were excluded from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
The effect of ten-day music therapy on anxiety levels of pregnant women | The music therapy application lasted for 10 days. Through study completion the final test of the a State and Trait Anxiety Inventory (STAI I-II) was performed with pregnant women.
  Pre-intervention, a personal information form and a State and Trait Anxiety Inventory (STAI I-II) (Oner and Le Compte, 1998) were used to assess the anxiety levels of pregnant women. The minimum score they will receive from the State and Trait Anxiety Inventory is 0, the maximum score is 80.
The effect of ten-day music therapy on stress levels of pregnant women | The music therapy application lasted for 10 days. Through study completion final test of the a Pregnancy Stress Rating Scale (PSRS) was performed with pregnant women.
  Pre-intervention, a Pregnancy Stress Rating Scale (Akin and Erbil, 2018) (PSRS) were used to assess the stress levels of pregnant women. The minimum score they will receive from the Pregnancy Stress Rating Scale is 0, the maximum is 144.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Ertaş, Master, Principal Investigator — Kutahya Health Sciences University; Neşe Çelik, Phd, Study Director — Eskisehir Osmangazi University
Locations (1):
- Kutahya Health Sciences University, Kütahya, Turkey (Türkiye)